CLINICAL TRIAL: NCT04816370
Title: Primary Sjögren's Syndrome Affects Female Genitalia and Sexual Functions: A Case Control Study
Brief Title: Effects of Primary Sjögren's Syndrome on Female Genitalia and Sexual Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Gozukucuk, Principal Investigator, Ankara Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: A1
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Primary Sjögren Syndrome
Keywords: primary Sjögren's Syndrome; vaginal atrophy; sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pSS group (Experimental): primary Sjögren's syndrome group
  Interventions: Diagnostic Test: FSFI
- Control Group (Experimental): Control group
  Interventions: Diagnostic Test: FSFI
- pSS Premenopausal (Experimental): primary Sjögren's syndrome premenopausal patients
  Interventions: Diagnostic Test: FSFI
- pSS Postmenopausal (Experimental): primary Sjögren's syndrome postmenopausal patients
  Interventions: Diagnostic Test: FSFI

INTERVENTIONS:
Diagnostic Test: FSFI — 2 group and 2 subgroup

SUMMARY:
A total of 68 women with pSS and 135 healthy female patients were included in the study. All women in the study and control groups were evaluated gynecologically, and genital findings during the examination and variables related to pSS were recorded. Women's sexual functions were evaluated with the Female Sexual Function Index (FSFI) and quality of life was evaluated using the Health Status Questionnaire-Short Form 36.

DETAILED DESCRIPTION:
This prospective, single-center, cross-sectional case control study will include a total of 68 women with pSS who presented to the rheumatology outpatient clinic of a tertiary care hospital and 135 healthy females who presented to the gynecology outpatient clinic for reasons other than sexual dysfunction and had similar age and menopausal status to the pSS group. The diagnosis of pSS was made according to the American-European Consensus Group criteria. Age, gravity, parity, body mass index (BMI), education status, smoking status, menarche age, and menopausal status and duration will be recorded for all participants. Disease duration, serum C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), anti-nuclear antibody (ANA) positivity, extractable nuclear antigen antibodies panel, extraglandular involvement and salivary gland pathologies were recorded. Disease-related variables (activity and function data, etc.), European League Against Rheumatism (EULAR) Sjögren's Syndrome Patient Reported Index (ESSPRI), EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI), Clinical Disease Activity Index (CDAI), Disease Activity Score 28 (DAS28), Health Assessment Questionnaire (HAQ), Visual Analog Scale-Pain (VAS-Pain) and fatigue scores and medicines used for pSS will be evaluated and recorded only in the pSS group. A gynecological examination will be performed in the lithotomy position in all participants in both groups by the same gynecologist with at least 15 years of professional experience. In order to determine vaginal atrophy, shrinkage and thinning of the mucosa, loss of rugae in the vagina and introitus stenosis are taken into consideration. The reduction of subcutaneous fat in the labia majora is evaluated as labial atrophy, and contraction in size and even retraction of the clitoral prepuce is interpreted as clitoral atrophy. Pain sensation on speculum examination will be assessed by VAS (rated from 0 to 10). Vaginal culture and cervico-vaginal smear will be analyzed, and the findings will be recorded.

Women aged over 20 and under 70 years will be included in the study. Pregnant patients and those with known hepatic, renal, interstitial lung, gynecological oncological diseases, psychiatric disorders, and communication impairment will be excluded from the study. The Female Sexual Function Index (FSFI), Health Status Questionnaire [Short Form (SF)-36], and Hospital Depression and Anxiety Scale (HADS) will be administered to the women in both groups, and their scores were recorded. The data obtained from the study and control groups will be compared. The patients in the pSS group and healthy controls will be further divided into two subgroups according to their menopause status, and statistical comparisons will also be undertaken between these subgroups. A multivariate linear regression analysis will be performed, and the correlation of sexual function with other parameters is examined.

ELIGIBILITY:
Inclusion Criteria:

Clinical Diagnosis of pSS healthy females who presented to the gynecology outpatient clinic for reasons other than sexual dysfunction -

Exclusion Criteria:

Pregnancy hepatic, renal, interstitial lung, gynecological oncological diseases, psychiatric disorders communication impairment

-

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Sexual Function | 1 day
  The sexual functions of women participating in the study were evaluated in six subdomains, arousal, desire, lubrication, orgasm, pain, and satisfaction.Higher scores demonstrate preferable sexual function. The total score is obtained by adding the scores of six-subdomains

CONTACTS AND LOCATIONS:
Overall Officials: Murat Gözüküçük, Principal Investigator — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Education Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maddali Bongi S, Del Rosso A, Orlandi M, Matucci-Cerinic M. Gynaecological symptoms and sexual disability in women with primary Sjogren's syndrome and sicca syndrome. Clin Exp Rheumatol. 2013 Sep-Oct;31(5):683-90. Epub 2013 May 27. PMID 23710558
- [Result] McCoy SS, Sampene E, Baer AN. Association of Sjogren's Syndrome With Reduced Lifetime Sex Hormone Exposure: A Case-Control Study. Arthritis Care Res (Hoboken). 2020 Sep;72(9):1315-1322. doi: 10.1002/acr.24014. PMID 31233285